CLINICAL TRIAL: NCT05166941
Title: In Psychiatric Nursing Education; The Effect of Creative Drama Method Based on Travelbee's "Human to Human Relationship" Theory on Developing Anxiety, Empathy and Communication Skills
Brief Title: THE EFFECT OF CREATIVE DRAMA ON THE DEVELOPMENT OF ANXIETY, EMPATHY AND COMMUNICATION SKILLS IN NURSING EDUCATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Günseli Uzunhasanoğlu, PhD student, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Ankara YBU-SBF-GU-01
Record Dates: First submitted 2021-12-12; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Psychiatric Nursing
Keywords: psychiatric nursing ,creative drama, empathy, Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: it was planned in a quantitative design as a randomized controlled intervention study and in a mixed method in qualitative design in order to examine students' views on the method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): It is a closed group in which the training program is implemented.
  Interventions: Behavioral: creative drama
- Control Group (No Intervention): No training program was applied to this group.

INTERVENTIONS:
Behavioral: creative drama — In the training program, a total of six games were played about the experiences of psychiatric patients. The program was designed to be two game per week for four weeks.
  Arms: Experimental group

SUMMARY:
This work; The aim of this study is to determine the effect of the education program, which was created with the creative drama method based on Travelbee's "human-to-human relationship" theory, on the teaching and practice of mental health and psychiatric nursing course, on reducing the anxiety of students and improving their empathy and communication skills.

DETAILED DESCRIPTION:
In psychiatric nursing education; It is known that classical education methods are not sufficient to reduce students' anxiety and stigma, and to strengthen communication and empathy. For this reason, there is a need for training methods that will increase in-depth learning and communication skills and empathy in the field. In this research, the creative drama education method was arranged in accordance with the requirements of mental health and psychiatric nursing education and a training program was developed. Within the scope of the research, this training program was applied to the students who completed the theoretical education of psychiatric nursing. In order to measure the effectiveness of the research training program, it was planned in a quantitative design as a randomized controlled intervention study and in a mixed method in qualitative design in order to examine students' views on the method.

ELIGIBILITY:
Inclusion Criteria:

* Being residing in the city center of Ankara Volunteering to participate in the research, Being a 4th year nursing student and having completed the Mental Health and Diseases Nursing course, Lack of clinical experience in communicating with individuals with mental illness (Health Vocational High School graduate), Not having received training in communicating with individuals with mental illness before (students repeating a grade).

Not having been diagnosed with any mental illness No mental illness in first degree relatives

Exclusion Criteria:

* Living outside the city center of Ankara To fill in the research data collection forms incompletely, Not completing the creative drama education based on human-human relationship theory, Refusal to participate in the research Not meeting the criteria for inclusion in the research

Ages: 21 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
The Numerical Rating Scale(NRS) | Eight weeks
  It was applied to the experimental and control groups to quantitatively measure the effectiveness of the training program.
Qualitative method, (focus group interview) | one weeks
  It was applied to evaluate the opinions and suggestions of the experimental group about the education program.

SECONDARY OUTCOMES:
Empathic Skill Scale - B | Eight weeks
  It was used to determine the level of empathic skills of the students at the end of the training program.
Communication Skills Assessment Scale | Eight weeks
  It was used to determine the level of communication skills of the students at the end of the education program.
State and Trait Anxiety Scale | Eight weeks
  It was used to determine the level of anxiety experienced by the students at the end of the education program.
semi-structured questionnaire | one weeks
  It was applied to evaluate the opinions and suggestions of the experimental group about the education program

CONTACTS AND LOCATIONS:
Overall Officials: günseli uzunhasanoğlu, Phd, Principal Investigator — Ankara Yildirim Beyazıt University; Birgul Ozkan, Phd, Study Director — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No